CLINICAL TRIAL: NCT03286803
Title: Comparison of Immunity Following Inactivated Poliovirus Vaccine Versus Fractional Dose Inactivated Poliovirus Vaccine: a Community Based Randomized Controlled Trial in Pakistan
Brief Title: Comparison of Immunity Following IPV Versus fIPV: a Community Based Randomized Controlled Trial in Pakistan
Acronym: CODI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Ali Faisal Saleem, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4624-Ped-ERC-17
Record Dates: First submitted 2017-09-11; First posted 2017-09-18 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Poliovirus Vaccine, Inactivated; Poliomyelitis; Immunization; Infection
MeSH Terms: conditions — Poliomyelitis; Infections | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Intervention Model Description: This will be a four arms randomized controlled trial. Arms 1 and 2 will randomize children aged 14 weeks old into either full dose or fractional dose IPV and arms 3 and 4 will randomize children aged 9 months old into either full dose or fractional dose IPV
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Inactivated Poliovirus vaccine
  Interventions: Biological: Inactivated Poliovirus vaccine
- Arm B (Active Comparator): fractional dose inactivated poliovirus vaccine
  Interventions: Biological: Inactivated Poliovirus vaccine
- Arm C (Experimental): inactivated poliovirus vaccine
  Interventions: Biological: Inactivated Poliovirus vaccine
- Arm D (Active Comparator): fractional dose inactivated poliovirus vaccine
  Interventions: Biological: Inactivated Poliovirus vaccine

INTERVENTIONS:
Biological: Inactivated Poliovirus vaccine — we will administer either full dose (0.5ml) or fractional dose (0.1ml) of inactivated poliovirus vaccine
  Other Names: fractional dose Inactivated Poliovirus vaccine

SUMMARY:
This study will be conducted in four low-income areas of Bin Qasim Town Karachi. This will be a community based randomized control trial of 21 months duration. The trial will include four arms; arm A and B will enroll children age 14-18 weeks and randomize them to either full dose IPV (0.5ml) or fractional IPV (0.1ml). Arms C and D will enroll children at 9 months of age and randomize them to either fractional or full dose IPV.

Children aged 14 weeks for arms A and B and 9 months for arms C and D living in the selected communities of Bin qasim Town Karachi who have not received IPV vaccine during routine immunization for arms A and B and who have documentary evidence of receiving IPV vaccine at 14 weeks of age for arms C and D will be eligible for enrollment.

The investigators will exclude children who are found acutely ill or those requiring emergent medical care/hospitalization at the time of enrollment.

The investigators will use the Demographic Surveillance System (DSS) in the four study areas to identify the households with eligible children. The children of the parents who agree to participate in the study will be screened for eligibility by the trained research associates. After randomization into four different arms, the study trained research vaccinators will administer the IPV or fIPV as per randomization. Children will be observed in the center for 30 minutes after vaccination before leaving for home. Parents/guardians of all the participants will also be requested to immediately report any adverse effect occurring later.

This study will be conducted in compliance with this protocol, GCP guidelines and all applicable international and local regulatory requirements. The study has approval by the Ethical Review Committee of the Aga Khan University (AKU), the National Bioethics Committee of Pakistan, and ethical approval at WHO/Headquarters in Geneva. All study procedures will be conducted in AKU's field research sites from where subjects will be recruited. The Clinical Trials Unit (CTU) of AKU will be engaged in providing support for specific study procedures conducted at CTU such as randomization, management of vaccines (storage, dispensing and incineration), and other responsibilities agreed in writing.

Adverse events following vaccine administration will be monitored and all serius adverse events will be reported within 24 hours to WHO, DSMB and AKU IRB. All the vaccines used are licensed in Pakistan and in routine use.

DETAILED DESCRIPTION:
Background In April 2016, there was globally synchronized switch from tOPV to bivalent OPV (bOPV). The Strategic Advisory Group of Experts on immunization (SAGE) from WHO endorsed the use of IPV in routine immunization globally.(1, 2) However, the IPV introduction pose challenges. The biggest challenge is sustain delivery and availability of IPV not only to the countries with endemic and periodic epidemic for polio disease but also for the countries at risk. Previous research demonstrate that fractional dose of IPV (fIPV) is as efficacious as IPV in children received OPV in their routine immunization.(3, 4) Many countries are in the process of introducing two doses of fIPV in their routine immunization. Pakistan is still one of the two remaining polio endemic countries. There has been gradual decline of wild polio virus 1 cases in 2016 (2014, 306 cases; 2015, 54 cases and 2016, 15 cases as of October 15). This decline is mainly because of strengthening routine immunization, introduction of bOPV and IPV in national polio campaigns. The data on PV2 seroconversion after the introduction of one or two doses of fIPV post bOPV introduction is lacking. There is no data on how long the PV2 serum immunity last. The current study focuses to assess seroconversion for PV2 induced by one and two dose schedule with IPV and compare to fIPV. The investigators also aim to assess the decline in titer within 12 months following second IPV dose and compare the decline between IPV and fIPV schedules.

Study Objectives

* To compare the immunogenicity and seroconversion of PV2 induced by of two doses IPV versus two doses of fractional IPV administered at 14 weeks and 9 months of age.
* To compare the immunogenicity of single dose IPV versus single dose fractional IPV administered at 14 weeks of age.
* To assess the decline in titer within 12 months following IPV compare the decline between IPV and fIPV schedule Methodology Description of the study setting and population Karachi is a large city with five districts and eighteen towns. This study will be conducted in four low-income areas in and around Karachi (4 peri-urban, contiguous coastal villages outside Karachi) located about half hour driving distance from AKU where the Aga Khan University's Department of Paediatrics and Child Health has well-established demographic surveillance, which captures all pregnancies and new births in the area.

Study design This will be a community based randomized control trial. Sample size Assuming 90% of immune response at 21 months of age after administration of two full doses of IPV, 80% power to detect the difference of 15% between arms, 5% level of significance and 10% of drop outs, the required minimum sample size will be 500 (125 in each arm).

Recruitment of the participants, study procedures and administration of informed consent

The investigators will use the Demographic Surveillance System (DSS) in the four study areas to identify the households with eligible children. The lists of these households with complete address will be retrieved from the DSS. Team of community health workers (CHWs) will visit eligible households and will explain the study to the mother/father or any legal guardian of the child. The children of the parents who agree to participate in the study will be screened for eligibility by the trained research associates. The parents of the children found eligible to be enrolled will be asked for the written informed consent. Eligible children will be enrolled if their parents or legal guardian provide the written informed consent. Special request permission will be obtained regarding following procedures:

1. To perform four blood draws of 2 ml each if the children is randomized to arm A or B and three blood draws if the child is randomized to arm C and D.

   (Maximum of two attempts for a blood draw will be performed)
2. To receive one additional IPV dose at 9 months if the child is randomized to arm A and either a single or two factional doses of IPV (1/5th of the normal dose) if the child is randomized to arm B or D.

Randomization Clinical Trial Unit (CTU) of the Aga khan University will be asked to generate two different lists of randomization using individual randomization technique. List 1 will be used for the randomization of children aged 14 weeks and they will be either randomized to arm A or B. List 2 will be used for the randomization of children aged 9 months and they will be either randomized to arm C or D.

Sample collection and analysis The investigators will collect 2 ml of venous blood at enrollment before the randomization and then at different follow up visits. Blood sample will be immediately centrifuged at the centers and sent to the central infectious disease research laboratory (IDRL) at Aga Khan University campus in Karachi for storage. The blood samples will be shipped to the Centers for Disease Control and Prevention in Atlanta, USA (CDC), and tested for presence of poliovirus neutralizing antibodies using neutralization assays. Any remaining sera will be destroyed after the assays are carried out.

Seropositivity is defined as reciprocal titers of poliovirus neutralizing antibodies >8; seroconversion is defined as the change from seronegative to seropositive (from reciprocal titer of <8 to >8); and boosting is defined as >4-fold increase in titers. In this study, "immune response" combines both boosting and seroconversion. The analysis of immune response will be restricted to infants with a baseline serological titer of < 362 to ensure that a 4-fold boosting response could be achieved since the highest titer tested will be 1:1,448. In addition, data on structured case report forms will be obtained in first visit (socio-demographic and anthropometric data), and at each subsequent visits.

CRF (Case Report Form): This brief questionnaire will include information on gender, age, weight, length, randomization, maternal education, and information on routine immunization of the child.

Data collection procedure Data will be collected by trained research assistants and vaccinators complying with Good Clinical Practice (GCP) standards. At enrollment each study subject will be assigned a unique identification number and all the subsequent questionnaires will be anonymized. This number will be used for future identification. Data will be collected using pre-designed and pilot tested questionnaires.

Monitoring and safety This study will be conducted in compliance with this protocol, GCP guidelines and all applicable international and local regulatory requirements. The study will require approval by the Ethical Review Committee of the Aga Khan University (AKU), the National Bioethics Committee of Pakistan, and ethical approval at WHO/Headquarters in Geneva. All study procedures will be conducted in AKU's field research sites from where subjects will be recruited. The Clinical Trials Unit (CTU) of AKU will be engaged in providing support for specific study procedures conducted at CTU such as randomization, management of vaccines (storage, dispensing and incineration), and other responsibilities agreed in writing.

Adverse events following vaccine administration will be monitored and all serius adverse events will be reported within 24 hours to WHO, DSMB, AKU online adverse drugs reporting (ADR), and AKU online medical incident reporting. Vaccines will be stored according to cold chain requirements, and detailed inventory logs will be maintained at the field sites and at the Clinical Trial Unit. There are no placebos used in this study. All the vaccines used are licensed in Pakistan and in routine use.

Specification of the safety parameters:

All participants will be informed to contact the study primary investigators or study physicians at the primary care area clinics if the child requires medical care. Should a serious illness arise requiring a physician visit or hospitalization, parents will receive instructions on who to contact. In the unforeseen instance of serious adverse events after routine immunization, free transport and hospital referral to an Aga Khan University Hospital will be arranged as well as provision of cost of care during hospital stay.

Study duration This will be an twenty one month study, starting in Aug, 2017.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 14 weeks for arms A and B and 9 months for arms C and D living in four peri-urban slums of Bin Qasim Town, Karachi (Rehri Goth, Bhains Colony, Ali Akber Shah, Ibrahim Hydri) who have not received IPV vaccine during routine immunization for arms A and B and who have documentary evidence of receiving IPV vaccine at 14 weeks of age for arms C and D.

Exclusion Criteria:

* Child found acutely ill at the time of enrolment and requiring emergent medical care/hospitalization
* Parents planning to shift out of the four communities during the study time (at least 18 months for arms A and B, and 1 year for arms C and D)
* Refusal of blood testing
* Already enrolled in any other clinical trial

Ages: 14 Weeks to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
sero-conversion defined as the change from seronegative to seropositive (from reciprocal titer of <8 to >8) | 14 weeks to 10 months of age and 9 months to 10 months
  The difference in seroconversion at 10 months of age between two full dose IPV versus two fractional dose IPV administered at 14 weeks and 9 months of age.

SECONDARY OUTCOMES:
Immune response defined as the combination of both seroconversion and boosting (defined as >4-fold increase in titers) | 14 weeks to 18 weeks, 9 months, 10 months and 21 months
  Comparison of the immune response at across different study arms at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Ali Saleem, Principal Investigator — Aga Khan University
Locations (1):
- Rehri goth, Ibrahim Hyderi, Ali Akbar Shah, and Bhens Colony, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
We will share aggregate data to the other researchers.

REFERENCES:
- [Derived] Saleem AF, Parkar S, Zehra SM, Kazi Z, Pethani A, Zhang Y, Mainou BA, Cavestany RL, Macklin G, Jeyaseelan V, Mach O. Two-Year Duration of Immunity of Inactivated Poliovirus Vaccine: A Follow-up Study in Pakistan in 2020. J Infect Dis. 2024 Jan 12;229(1):39-42. doi: 10.1093/infdis/jiad237. PMID 37368349
- [Derived] Saleem AF, Mach O, Yousafzai MT, Kazi Z, Baig A, Sajid M, Jeyaseelan V, Sutter RW, Zaidi AKM. One-Year Decline of Poliovirus Antibodies Following Fractional-Dose Inactivated Poliovirus Vaccine. J Infect Dis. 2021 Apr 8;223(7):1214-1221. doi: 10.1093/infdis/jiaa504. PMID 32798224